CLINICAL TRIAL: NCT03141606
Title: Left Atrial Volume as Predictor for Arrhythmic Events and CRT Response
Acronym: iLAV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Borgo Trento - Verona (Other)
Responsible Party: Principal Investigator, Dr. Giovanni Morani, MD, Ospedale Borgo Trento - Verona
Other Study IDs: 20140002277
Record Dates: First submitted 2017-04-26; First posted 2017-05-05 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Left Atrial Volume

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Left atrial volume role for CRT response and for arrhythmic events (VT/VF/AT/AF) onset

ELIGIBILITY:
Inclusion Criteria:

* Patient with left ventricular ejection fraction ≤ 35%, II, III or IV NYHA Class, even if optimal medical therapy.
* Patients with standard indication to CRT according current guideline, sinus rhythm at implantation, LBBB and QRS duration >= 120 ms
* Patients who will undergo to a new CRT-defibrillator system implantation
* Patients who are able to understand and sign the informed consent
* Patients who are able to attend all required follow-up visits at the study centerfor 24 months

Exclusion Criteria:

* Age < 18 years
* Women who are pregnant or who are planning to become pregnant
* Patients with permanent Atrial Fibrillation or persistent Atrial Fibrillation in the 90 days preceding the implantation
* Patients with organic mitral valve disease
* Patients with prosthetic heart valves
* Patients who will undergo to upgrading from other devices (PM or ICD) to CRT, heart transplantation, patients with CRT devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with cardiac resynchronization therapy defirbillator devices and who meet the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Cardiac remodelling | 6 months
  Evaluation of function and volume of left atrium (by means of echocardiographic measures) in terms of cardiac remodelling (at least 15% reduction in LVESV).
CRT Predictor Index | 6 months
  Identification of left atrial index predicting CRT response

SECONDARY OUTCOMES:
Clinical benefit | 12 months
  Left atrial volume/function in terms of clinical benefit
  * Clinical Composite Score evaluation
  * QoL evaluation
Cardiac remodelling | 6 months
  Left atrial volume/function in terms of cardiac remodelling
  * LVEF
  * LVESV/LVEF
Atrial arrhythmias | 24 months
  Left atrial volume/function role in terms of:
  * atrial arrhythmias onset
  * Atrial arrhythmias burden
Ventricular arrhythmias | 24 months
  Left atrial volume/function in terms of:
  * ventricular arrhythmias onset
  * ventricular arrhythmias burden

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - G. Panico Hospital, Tricase, Italy/Lecce
  - Borgo Trento Hospital, Verona